CLINICAL TRIAL: NCT01229488
Title: System for Ocular Oxygen Measurement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: I withdrew from this study
Sponsor: Indiana University (Other)
Responsible Party: Joseph A. Bonanno, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 1006001474 IND
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Normal
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- No Arms (No Intervention): Project was withdrawn before starting
  Interventions: Device: Intervention

INTERVENTIONS:
Device: Intervention — Project was withdrawn before starting. There were no interventions

SUMMARY:
The purpose of this study is to demonstrate the ability of the OcuMetrics system to measure oxygen on the surface of the eye. Oxygen is important to the health of the cornea. The proposed instrument will take advantage of phosphorescent dyes that are sensitive to oxygen concentrations to monitor oxygen concentrations on the surface of the eye. This will have obvious applications in eye research and contact lens testing.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* contact lens wear in last 6 weeks
* Use of topical drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
oxygen tension measurement by new device is comparable with gold standard, but less variable and faster. | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Optometry, Bloomington, Indiana, United States